CLINICAL TRIAL: NCT00922974
Title: Phase II/III Study of Image-Guided Radiosurgery/SBRT for Localized Spine Metastasis
Brief Title: Image-Guided Radiosurgery or Stereotactic Body Radiation Therapy in Treating Patients With Localized Spine Metastasis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RTOG-0631; CDR0000646803; NCI-2009-01687 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2009-06-17; First posted 2009-06-18 (Estimated); Results first posted 2019-05-16 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2021-04

CONDITIONS: Metastatic Cancer; Pain
Keywords: spinal bone metastases; pain
MeSH Terms: conditions — Neoplasm Metastasis; Pain | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Radiosurgery/SBRT (Experimental)
  Interventions: Radiation: Radiosurgery/SBRT
- External Beam Radiation Therapy (Active Comparator)
  Interventions: Radiation: External beam radiation therapy

INTERVENTIONS:
Radiation: External beam radiation therapy — Single fraction dose of 8 Gy external beam radiation therapy
  Other Names: EBRT
  Arms: External Beam Radiation Therapy
Radiation: Radiosurgery/SBRT — Single fraction dose image-guided radiosurgery / stereotactic body radiotherapy (SBRT). The phase II component uses 16 Gy. The phase III component allows 16 or 18 Gy as preferred by the treating physician.
  Other Names: stereotactic body radiotherapy; SRS; stereotactic radiosurgery
  Arms: Radiosurgery/SBRT

SUMMARY:
RATIONALE: Specialized radiation therapy that delivers a high dose of radiation directly to the tumor may kill more tumor cells and cause less damage to normal tissue.

PURPOSE: This randomized phase II/III trial is studying how well image-guided radiosurgery or stereotactic body radiation therapy works and compares it to external-beam radiation therapy in treating patients with localized spine metastasis.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the feasibility of successfully delivering image-guided radiosurgery or stereotactic body radiotherapy (SBRT) in patients with spine metastases in a cooperative group setting. (Phase II)
* Determine whether image-guided radiosurgery or SBRT (single dose of 16 Gy) improves pain control as measured by the 11-point Numerical Rating Pain Scale (NRPS) compared to conventional external beam radiotherapy (single dose of 8 Gy). (Phase III)

Secondary

* Determine whether image-guided radiosurgery or SBRT improves the rapidity of pain response and increases the duration of pain response at the treated site(s) compared to conventional external beam radiotherapy, as measured by the NRPS. (Phase III)
* Compare adverse events associated with these treatment regimens, as measured by NCI CTCAE v3.0 criteria. (Phase III)
* Evaluate the long-term effects (24 months) of image-guided radiosurgery or SBRT on the vertebral bone (e.g., compression fracture) and the spinal cord, as measured by MRI. (Phase III)

DETAILS:

This is a multicenter, phase II study followed by a randomized phase III study. Patients enrolled in the phase III portion are stratified according to the number of spine metastases to be treated (1 vs 2-3) and the type of tumor (radioresistant [including soft tissue sarcomas, melanomas, and renal cell carcinomas] vs other).

Phase II patients undergo MRI of the treated spine at baseline and at 3 months; phase III patients undergo MRI at baseline and at 3, 6, 12, and 24 months. Patients enrolled in the phase III portion also complete the Numerical Rating Pain Scale at baseline, at 1, 2, and 3 weeks after randomization, and at 1, 3, 6, 12, and 24 months. Patients are followed after completion of study treatment.

ELIGIBILITY:
Inclusion Criteria:

1. The patient must have localized spine metastasis from the C1 to L5 levels by a screening imaging study [bone scan, positron emission tomography (PET), computerized tomography (CT), or magnetic resonance imaging (MRI)] (a solitary spine metastasis; two separate spine levels; or up to 3 separate sites [e.g., C5, T5-6, and T12] are permitted.) Each of the separate sites may have a maximal involvement of 2 contiguous vertebral bodies. Patients can have other visceral metastasis, and radioresistant tumors (including soft tissue sarcomas, melanomas, and renal cell carcinomas) are eligible. See Figure 1 in Section 3.1.1. of the protocol for a depiction of eligible metastatic lesions: 1) a solitary spine metastasis; 2) two contiguous spine levels involved; or 3) a maximum of 3 separate sites. Each of the separate sites may have a maximal involvement of 2 contiguous vertebral bodies. Epidural compression (arrow) is eligible when there is a ≥ 3 mm gap between the spinal cord and the edge of the epidural lesion (see #10). A paraspinal mass ≤ 5 cm is allowed (see #11).

   * There can be multiple small metastatic lesions shown in other vertebral bodies as shown in referenced diagram. The metastatic lesion of each spine should be less than 20% of the vertebral body as opposed to the diffuse vertebral involvement. These small lesions are often seen in the MRI even when bone scan or PET was negative. Most of these lesions are not clinically required to be treated and are therefore not included in the target volume of this protocol. Only the painful spine (pain score≥ 5) is to be treated .
2. Zubrod Performance Status 0-2;
3. Age ≥ 18;
4. History/physical examination within 2 weeks prior to registration;
5. Negative serum pregnancy test within 2 weeks prior to registration for women of childbearing potential;
6. Women of childbearing potential and male participants who are sexually active must agree to use a medically effective means of birth control;
7. MRI (contrast is not required but strongly recommended) of the involved spine within 4 weeks prior to registration to determine the extent of the spine involvement; an MRI is required as it is superior to a CT scan in delineating the spinal cord as well as identifying an epidural or paraspinal soft tissue component. Note: If an MRI was done as a screening imaging study for eligibility (see Section -1), the MRI can be used as the required MRI for treatment planning.
8. Numerical Rating Pain Scale within 1 week prior to registration; the patient must have a score on the Scale of ≥ 5 for at least one of the planned sites for spine radiosurgery. Documentation of the patient's initial pain score is required. Patients taking medication for pain at the time of registration are eligible.
9. Neurological examination within 1 week prior to registration to rule out rapid neurologic decline; see Appendix III for the standardized neurological examination. Patients with mild to moderate neurological signs are eligible. These neurological signs include radiculopathy, dermatomal sensory change, and muscle strength of involved extremity 4/5 (lower extremity for ambulation or upper extremity for raising arms and/or arm function).
10. Patients with epidural compression are eligible provided that there is a ≥ 3 mm gap between the spinal cord and the edge of the epidural lesion.
11. Patients with a paraspinal mass ≤ 5 cm in the greatest dimension and that is contiguous with spine metastasis are eligible.
12. Patients must provide study specific informed consent prior to study entry.

Exclusion Criteria:

1. Histologies of myeloma or lymphoma;
2. Non-ambulatory patients;
3. Spine instability due to a compression fracture;
4. > 50% loss of vertebral body height;
5. Frank spinal cord compression or displacement or epidural compression within 3 mm of the spinal cord;
6. Patients with rapid neurologic decline;
7. Bony retropulsion causing neurologic abnormality;
8. Prior radiation to the index spine;
9. Patients for whom an MRI of the spine is medically contraindicated;
10. Patients allergic to contrast dye used in MRIs or CT scans or who cannot be premedicated for the use of contrast dye.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 399 (Actual)
Dates: Start 2009-11 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2020-04-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Ryu, MD, Principal Investigator — Josephine Ford Cancer Center
Locations (38):
- United States (34):
  - University of Colorado Cancer Center at UC Health Sciences Center, Aurora, Colorado
  - Penrose Cancer Center at Penrose Hospital, Colorado Springs, Colorado
  - George Bray Cancer Center at the Hospital of Central Connecticut - New Britain Campus, New Britain, Connecticut
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Baptist Cancer Institute - Jacksonville, Jacksonville, Florida
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Cancer Center at Ball Memorial Hospital, Muncie, Indiana
  - Lucille P. Markey Cancer Center at University of Kentucky, Lexington, Kentucky
  - James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - St. Agnes Hospital Cancer Center, Baltimore, Maryland
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - Butterworth Hospital at Spectrum Health, Grand Rapids, Michigan
  - William Beaumont Hospital - Royal Oak Campus, Royal Oak, Michigan
  - Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri
  - Billings Clinic - Downtown, Billings, Montana
  - Nebraska Medical Center, Omaha, Nebraska
  - Payson Center for Cancer Care at Concord Hospital, Concord, New Hampshire
  - Seacoast Cancer Center at Wentworth - Douglass Hospital, Dover, New Hampshire
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Capital Health Regional Cancer Center, Pennington, New Jersey
  - Stony Brook University Cancer Center, Stony Brook, New York
  - Summa Center for Cancer Care at Akron City Hospital, Akron, Ohio
  - Arthur G. James Cancer Hospital and Richard J. Solove Research Institute at Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Penn State Hershey Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Kimmel Cancer Center at Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - UPMC - Shadyside, Pittsburgh, Pennsylvania
  - UPMC Cancer Center at UPMC Presbyterian, Pittsburgh, Pennsylvania
  - Lankenau Cancer Center at Lankenau Hospital, Wynnewood, Pennsylvania
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Huntsman Cancer Institute at University of Utah, Salt Lake City, Utah
  - University of Wisconsin Paul P. Carbone Comprehensive Cancer Center, Madison, Wisconsin
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin
  - All Saints Cancer Center at Wheaton Franciscan Healthcare, Racine, Wisconsin
- Canada (3):
  - Ottawa Hospital Regional Cancer Centre - General Campus, Ottawa, Ontario
  - Hopital Notre-Dame du CHUM, Montreal, Quebec
  - McGill Cancer Centre at McGill University, Montreal, Quebec
- Tel-Aviv Sourasky Medical Center, Tel Aviv, Israel

REFERENCES:
- [Result] Ryu S, Pugh SL, Gerszten PC, Yin FF, Timmerman RD, Hitchcock YJ, Movsas B, Kanner AA, Berk LB, Followill DS, Kachnic LA. RTOG 0631 phase 2/3 study of image guided stereotactic radiosurgery for localized (1-3) spine metastases: phase 2 results. Pract Radiat Oncol. 2014 Mar-Apr;4(2):76-81. doi: 10.1016/j.prro.2013.05.001. Epub 2013 Jun 4. PMID 24890347
- [Derived] Ryu S, Deshmukh S, Timmerman RD, Movsas B, Gerszten P, Yin FF, Dicker A, Abraham CD, Zhong J, Shiao SL, Tuli R, Desai A, Mell LK, Iyengar P, Hitchcock YJ, Allen AM, Burton S, Brown D, Sharp HJ, Dunlap NE, Siddiqui MS, Chen TH, Pugh SL, Kachnic LA. Stereotactic Radiosurgery vs Conventional Radiotherapy for Localized Vertebral Metastases of the Spine: Phase 3 Results of NRG Oncology/RTOG 0631 Randomized Clinical Trial. JAMA Oncol. 2023 Jun 1;9(6):800-807. doi: 10.1001/jamaoncol.2023.0356. PMID 37079324
- Available data/document: Individual Participant Data Set: NCT00922974 — https://nctn-data-archive.nci.nih.gov/ — Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive.

RESULTS

PARTICIPANT FLOW:
Period: Phase II Component
Arm/Group | Radiosurgery/SBRT | External Beam Radiation Therapy
Started | 46 | 0
Eligible | 44 | 0
Eligible and Started Treatment | 39 | 0
Eligible, Treated, Adverse Event Data (Eligible, started protocol treatment, and has adverse event data) | 34 | 0
Completed (Subjects contributing any data to analysis are considered to have completed the study) | 39 (These subjects do not participate in the phase III component.) | 0
Not Completed | 7 | 0
Not completed — Protocol Violation | 2 | 0
Not completed — Not evaluable for treatment review | 5 | 0
Period: Phase III Component
Arm/Group | Radiosurgery/SBRT | External Beam Radiation Therapy
Started | 217 (The phase III component accrues new subjects; these are not continuing phase II subjects.) | 136
Eligible | 209 | 130
Eligible With 3 mo. NRPS Data (All eligible randomized patients with both baseline and 3 month NRPS scores) | 139 | 76
Eligible With 3 mo. FACT-G Data (Eligible and QOL consented patients with both baseline and follow up 3 month FACT-G total Score) | 87 | 58
Eligible With Adverse Event Data | 202 | 117
Eligible, Treated, Adverse Event Data (Eligible, started protocol treatment, and has adverse event data) | 148 | 83
Eligible and Consented to Quality of Life Participate in Quality of Life (QOL) Study Component | 152 | 100
Completed (Subjects contributing any data to analysis are considered to have completed the study) | 209 | 130
Not Completed | 8 | 6
Not completed — Protocol Violation | 8 | 6

BASELINE CHARACTERISTICS:
Population: Eligible registered patients
Groups:
- Radiosurgery/SBRT (Phase II): Single fraction dose image-guided radiosurgery / stereotactic body radiotherapy (SBRT). The phase II component uses 16 Gy.
- Radiosurgery/SBRT (Phase III): Single fraction dose image-guided radiosurgery / stereotactic body radiotherapy (SBRT). The phase III component allows 16 or 18 Gy as preferred by the treating physician.
- Total: Total of all reporting groups
Arm/Group | Radiosurgery/SBRT (Phase II) | Radiosurgery/SBRT (Phase III) | External Beam Radiation Therapy | Total
Number analyzed (Participants) | 44 | 209 | 130 | 383
Age, Continuous [Median (Full Range); unit: years] | 63 [25 to 89] | 63 [23 to 93] | 63 [32 to 91] | 63 [23 to 93]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 95 | 60 | 173
  Male | 26 | 114 | 70 | 210
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 10 | 7 | 20
  Not Hispanic or Latino | 40 | 194 | 118 | 352
  Unknown or Not Reported | 1 | 5 | 5 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 0 | 2
  Asian | 0 | 12 | 3 | 15
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Black or African American | 5 | 20 | 20 | 45
  White | 38 | 169 | 101 | 308
  More than one race | 0 | 1 | 1 | 2
  Unknown or Not Reported | 0 | 6 | 4 | 10
Zubrod performance status [Count of Participants; unit: Participants] — Measure Description: 0 - Asymptomatic; 1 - Symptomatic but completely ambulatory; 2 - Symptomatic, <50% in bed during the day; 3 - Symptomatic, >50% in bed, but not bedbound; 4 - Bedbound; 5 - Death
  Participants
    0 | 13 | 51 | 34 | 98
    1 | 25 | 112 | 83 | 220
    2 | 6 | 46 | 13 | 65
Baseline Numerical Rating Pain Scale (NRPS) [Median (Full Range); unit: units on a scale] — Eleven-point scale 0-10 with 0 indicating no pain and 10 indicating the worst pain imaginable.
  units on a scale | 7 [0 to 10] | 7 [5 to 10] | 7 [5 to 10] | 7 [0 to 10]
Number of Spine Metastases [Count of Participants; unit: Participants]
  1 | 36 | 160 | 100 | 296
  2-3 | 8 | 49 | 30 | 87
Location of Index Spine Metastasis [Count of Participants; unit: Participants] — The index site is the lesion with the highest baseline (day of radiosurgery) pain score. If multiple sites have the same baseline pain score, the index site is the most cephalad lesion.
  Participants
    C-1 to C-7 | 4 | 9 | 11 | 24
    T-1 to T-6 | 6 | 36 | 19 | 61
    T-7 to T-12 | 15 | 65 | 50 | 130
    L-1 to L-5 | 19 | 99 | 50 | 168
Location of Spine Metastasis #2 [Count of Participants; unit: Participants] — Population: Subjects who had a second metastasis
  Participants
    number analyzed (Participants) | 8 | 49 | 30 | 87
    C-1 to C-7 | 1 | 0 | 3 | 4
    T-1 to T-6 | 2 | 5 | 5 | 12
    T-7 to T-12 | 1 | 14 | 9 | 24
    L-1 to L-5 | 4 | 30 | 13 | 47
Location of Spine Metastasis #3 [Count of Participants; unit: Participants] — Population: Subjects who had a third metastasis
  Participants
    number analyzed (Participants) | 1 | 6 | 10 | 17
    T-1 to T-6 | 0 | 1 | 2 | 3
    T-7 to T-12 | 0 | 3 | 5 | 8
    L-1 to L-5 | 1 | 2 | 3 | 6
Taking Pain Medication [Count of Participants; unit: Participants]
  No | 2 | 28 | 15 | 45
  Yes | 42 | 181 | 115 | 338
Type of Tumor [Count of Participants; unit: Participants] — Population: This characteristic was not determined in the Phase II component.
  Participants
    number analyzed (Participants) | 0 | 209 | 130 | 339
    Radioresistant |  | 29 | 15 | 44
    Other |  | 180 | 115 | 295
Intended Radiosurgery/SBRT Dose [Count of Participants; unit: Participants]
  16 Gy | 44 | 115 | 76 | 235
  18 Gy | 0 | 94 | 54 | 148

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Receiving Radiosurgery/SBRT Per Protocol or With Minor Variation (Phase II)
Description: Treatment delivery was centrally reviewed by the study chair and medical physics co-chair. Success was defined as having a review of "per protocol" or "minor variation". A 70% success rate was required for continuation to the phase III component.
  * Target volume compliance in is defined as the following levels of target coverage in reference to dose volume:
    * Per protocol: ≥ 90%
    * Minor variation: 80%-90%
    * Major deviation: <80% of of dose volume.
  * Image-Guided Radiotherapy (IGRT) compliance is defined as the following differences in IGRT images between simulation/planning and treatment, as well as at the end of treatment:
    * Per protocol: <2 mm
    * Minor variation: 2mm - 3mm
    * Major deviation: > 3mm
Time Frame: The day of protocol treatment
Population: Patients enrolled in the phase II component who were eligible and had treatment review information.
Measure: Count of Participants; unit: Participants
Arm/Group | Radiosurgery/SBRT (Phase II)
Number analyzed (Participants) | 39
Participants
  Target volume | 39
  IGRT | 37

2. Primary Outcome: Percentage of Patients With Complete or Partial Pain Response at 3 Months (Phase III)
Description: Pain is measured by the Numerical Rating Pain Scale (NRPS) a numerical 11-point scale (0-10) with 0 = no pain, 1-4 = mild, 5-6 = moderate, and 7-10 = severe with 10 the worst pain imaginable. Pain response is calculated as 3 month score - baseline score with a positive value indicating increased pain and a negative value indicating decreased pain. Patients with complete or partial pain response as defined below are considered responders. The index site is the lesion with the highest baseline (day of radiosurgery) pain score. If multiple sites have the same baseline pain score, the index site is the most cephalad lesion.
  * Complete response: post-treatment pain score of 0 at the index site, no increase in narcotic pain medication, and no increase in pain score at the secondary treated site(s).
  * Partial response: post-treatment improvement of at least 3 points at the index site, no increase in narcotic pain medication, and no increase in pain score at the secondary treated site(s).
Time Frame: Baseline and 3 months
Population: Eligible participants randomized in the phase III component with both baseline and 3 month NRPS scores
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Radiosurgery/SBRT (Phase III) | External Beam Radiation Therapy
Number analyzed (Participants) | 139 | 76
percentage of participants | 40.3 [32 to 49] | 57.9 [46 to 69]
Statistical Analysis 1: Comparison: Radiosurgery/SBRT (Phase III) vs External Beam Radiation Therapy; Based on the one-sided exact binomial test with α=0.025 and a 2:1 randomization, 228 patients would be required to detect a 40% improvement in the response rate from 51% (external beam radiation therapy) to 70% (Radiosurgery/SBRT) with a statistical power of 0.80; Test type: Superiority; p = 0.99, Fisher Exact

3. Secondary Outcome: Percentage of Participants With Pain Response Through Two Years (Phase III)
Description: Pain is measured by the NRPS, a numerical 11-point scale from 0=no pain to 10=worst pain imaginable. Magnitude of pain response = post-baseline score - baseline score with a positive value indicating increased pain and a negative value indicating decreased pain. Pain response begins when a patient improves at least 3 points at the index site. (Although pain medication and pain response were part of the protocol definition of pain response, they were unable to be assessed accurately during weeks 1-3 and therefore were not included in the final definition used here.) Pain response time is defined as time from randomization to the date of pain response, last known follow-up (censored), or death (censored). Rates of participants with pain response are estimated using the Kaplan-Meier method. The distributions of pain response times are compared between the arms. Two-year rates are provided.
Time Frame: Baseline to two years. NRPS measured at baseline, 1, 2, and 3 weeks, 3, 6, 12, and 24 months.
Population: Eligible participants randomized in the phase III component with pain response data
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Radiosurgery/SBRT (Phase III) | External Beam Radiation Therapy
Number analyzed (Participants) | 209 | 130
percentage of participants | 19.2 [11.6 to 26.8] | 19.2 [9.6 to 28.7]
Statistical Analysis 1: Comparison: Radiosurgery/SBRT (Phase III) vs External Beam Radiation Therapy; Test type: Superiority; p = 0.38, Stratified log rank; One-sided significance level = 0.025; Hazard Ratio (HR) = 0.96, 95% CI 2-sided [0.72 to 1.27] — Reference level = Radiosurgery/SBRT

4. Secondary Outcome: Percentage of Participants With Pain Relapse Through Two Years (Phase III)
Description: Pain is measured by the NRPS, a numerical 11-point scale from 0=no pain to 10=worst pain imaginable. Amount of pain response = post-baseline score - baseline score with a positive value indicating increased pain and a negative value indicating decreased pain. Pain response begins when a patient improves at least 3 points at the index site. Pain response ends when when the pain score increases by 3 points (relapse). (Although pain medication and pain response were part of the protocol definition of pain response, they were unable to be assessed accurately during weeks 1-3 and therefore were not included in the final definition used here.) Pain relapse time is defined as time from randomization to the date of first failure, last known follow-up (censored), or death (censored). Rates of participants with pain relapse are estimated using the Kaplan-Meier method. The distributions of pain relapse times are compared between the arms. Two-year rates are provided.
Time Frame: Randomization to two years. NRPS measured at baseline, 1, 2, and 3 weeks, 3, 6, 12, and 24 months.
Population: Eligible participants randomized in the phase III component who experienced partial or complete pain response
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Radiosurgery/SBRT (Phase III) | External Beam Radiation Therapy
Number analyzed (Participants) | 140 | 80
percentage of participants | 91.7 [84.9 to 98.6] | 96.9 [92.6 to 100]
Statistical Analysis 1: Comparison: Radiosurgery/SBRT (Phase III) vs External Beam Radiation Therapy; Test type: Superiority; p = 0.29, Stratified log rank; One-sided significance level = 0.025; Hazard Ratio (HR) = 1.73, 95% CI 2-sided [0.24 to 12.8] — Significance level = Radiosurgery/SBRT

5. Secondary Outcome: Percentage of Patients With Adverse Events at 3 Months (Phase III)
Description: Common Terminology Criteria for Adverse Events (version 3.0) grades adverse event (AE) severity from 1=mild to 5=death. Summary data is provided in this outcome measure.; See Adverse Events Module for specific adverse event data.
Time Frame: Baseline to 3 months
Population: Eligible participants randomized in the phase III component with adverse event information
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Radiosurgery/SBRT (Phase III) | External Beam Radiation Therapy
Number analyzed (Participants) | 202 | 117
percentage of participants
  Treatment-related AE | 7.4 [3.8 to 11.0] | 7.7 [2.8 to 12.5]
  Any AE | 43.6 [36.7 to 50.0] | 36.7 [28.0 to 45.5]
Statistical Analysis 1: Comparison: Radiosurgery/SBRT (Phase III) vs External Beam Radiation Therapy; Percentage of patients with treatment-related adverse events; Test type: Superiority; p = 0.93, Chi-squared — Two-sided significance level = 0.05
Statistical Analysis 2: Comparison: Radiosurgery/SBRT (Phase III) vs External Beam Radiation Therapy; Percentage of patients with any adverse events; Test type: Superiority; p = 0.09, Chi-squared — Two-sided significance level = 0.05

6. Secondary Outcome: Percentage of Participants With a Vertebral Compression Fracture Through Two Years (Phase III)
Description: Failure is defined as a vertebral compression fracture. Failure time is defined as time from randomization to the date of first failure, last known follow-up (censored), or death without compression fracture (competing risk). Failure rates are estimated using the cumulative incidence method. The distributions of failure times are compared between the arms. Two-year rates are provided.
Time Frame: From randomization to two years.
Population: Eligible participants randomized in the phase III component
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Radiosurgery/SBRT (Phase III) | External Beam Radiation Therapy
Number analyzed (Participants) | 209 | 130
percentage of participants | 19.5 [14.3 to 25.3] | 21.6 [14.6 to 29.6]
Statistical Analysis 1: Comparison: Radiosurgery/SBRT (Phase III) vs External Beam Radiation Therapy; Test type: Superiority; p = 0.59, Gray's test — Two-sided significance level = 0.05

7. Secondary Outcome: Percentage of Participants With Spinal Cord Damage Through Two Years
Description: Failure is defined as spinal cord damage. Failure time is defined as time from randomization to the date of first failure, last known follow-up (censored), or death without compression fracture (competing risk). Failure rates are estimated using the cumulative incidence method. The distributions of failure times are compared between the arms. Two-year rates are provided.
Time Frame: From randomization to two years
Population: Eligible participants randomized in the phase III component
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Radiosurgery/SBRT (Phase III) | External Beam Radiation Therapy
Number analyzed (Participants) | 209 | 130
percentage of participants | 3.6 [1.6 to 6.9] | 1.7 [0.3 to 5.4]
Statistical Analysis 1: Comparison: Radiosurgery/SBRT (Phase III) vs External Beam Radiation Therapy; Test type: Superiority; p = 0.38, Gray's test — Two-sided significance level = 0.05

8. Secondary Outcome: Change in Functional Assessment of Cancer Therapy - General (FACT-G) Total Score at 3 Months (Phase III)
Description: The FACT-G is a validated 27-item measure in which a higher score represents higher quality of life (QOL). Physical, functional, social and emotional well-being subscale scores are added together to form the FACT-G total score. Responses range from 0=Not a lot to 4=Very much. Certain items must be reversed before being added, by subtracting the response from 4. Subscale items are added together, multiplied by the number of items in the subscale, then divided by the number of items answered to obtain subscale totals. Total score ranges from 0-108; physical, social and functional subscales from 0-28; emotional subscale from 0-24. Each subscale requires at least 50% of the items to be completed while the overall response rate must be greater than 80%. If items are missing the subscale scores can be prorated. Change at 3 months is calculated as 3 month score - baseline score with a positive change indicating improvement in QOL.
Time Frame: Baseline and 3 months
Population: Eligible patients randomized in the phase III component who consented to QOL having both baseline and 3 month FACT-G total score.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Radiosurgery/SBRT (Phase III) | External Beam Radiation Therapy
Number analyzed (Participants) | 87 | 58
score on a scale | 2.4 (16.0) | 5.2 (14.1)
Statistical Analysis 1: Comparison: Radiosurgery/SBRT (Phase III) vs External Beam Radiation Therapy; Assuming that the data are normally distributed, the two sample t-test assuming equal variances will be used to test the hypothesis at the one-sided 0.025 significance level. A mean difference of 7 points represents a clinically meaningful change (CMC). A difference of less than 7 points between the treatment arms will not be considered meaningful, even if it has statistical significance; Test type: Superiority; p = 0.28, t-test, 2 sided

9. Secondary Outcome: Change in Brief Pain Inventory (BPI) Worst Pain Score Through Two Years (Phase III)
Description: The Brief Pain Inventory Worst Pain score measures self-reported worst pain in the last week. Possible scores range from 0 (no pain) to 10 (worst pain imaginable), with higher scores indicating a worse outcome. Change is calculated as baseline score subtracted from post-baseline score with a positive change indicating more pain.
Time Frame: Baseline, 3, 6, 12, and 24 months
Population: Questionnaires were not completed by all eligible participants randomized in the phase III component who consented to QOL. Therefore, the number of participants reported below are the number with the relevant questions answered at baseline and the given time point on each arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Radiosurgery/SBRT (Phase III) | External Beam Radiation Therapy
Number analyzed (Participants) | 152 | 100
score on a scale
  3 months: number analyzed (Participants) | 80 | 49
  3 months | -1.9 (2.9) | -2.0 (3.3)
  6 months: number analyzed (Participants) | 43 | 27
  6 months | -2.3 (2.9) | -2.8 (2.9)
  12 months: number analyzed (Participants) | 35 | 29
  12 months | -2.2 (3.7) | -2.3 (2.9)
  24 months: number analyzed (Participants) | 25 | 12
  24 months | -1.4 (3.3) | -2.1 (3.5)
Statistical Analysis 1: Comparison: Radiosurgery/SBRT (Phase III) vs External Beam Radiation Therapy; A general linear mixed-effect model was run with BPI Worst Pain Score (baseline, 3, 6, 12, and 24 months) as the outcome of interest. Age, gender, race, Zubrod performance status, pain medication, tumor type, time, and treatment arm were the covariates considered in each model. Treatment Arm (External Beam Radiation Therapy vs. Radiosurgery/SBRT) is reported here; Test type: Superiority; p = 0.4313, Mixed Models Analysis; Each explanatory variable is reported separately. (Time and intercept estimates are not shown.)
Statistical Analysis 2: Comparison: Radiosurgery/SBRT (Phase III) vs External Beam Radiation Therapy; A general linear mixed-effect model was run with BPI Worst Pain Score (baseline, 3, 6, 12, and 24 months) as the outcome of interest. Age, gender, race, Zubrod performance status, pain medication, tumor type, time, and treatment arm were the covariates considered in each model. Age (< 63 years vs. ≥ 63 years) is reported here; Test type: Superiority; p = 0.8707, Mixed Models Analysis; Each explanatory variable is reported separately. (Time and intercept estimates are not shown.)
Statistical Analysis 3: Comparison: Radiosurgery/SBRT (Phase III) vs External Beam Radiation Therapy; A general linear mixed-effect model was run with BPI Worst Pain Score (baseline, 3, 6, 12, and 24 months) as the outcome of interest. Age, gender, race, Zubrod performance status, pain medication, tumor type, time, and treatment arm were the covariates considered in each model. Gender (female vs. male) is reported here; Test type: Superiority; p = 0.1549, Mixed Models Analysis; Each explanatory variable is reported separately. (Time and intercept estimates are not shown.)
Statistical Analysis 4: Comparison: Radiosurgery/SBRT (Phase III) vs External Beam Radiation Therapy; A general linear mixed-effect model was run with BPI Worst Pain Score (baseline, 3, 6, 12, and 24 months) as the outcome of interest. Age, gender, race, Zubrod performance status, pain medication, tumor type, time, and treatment arm were the covariates considered in each model. Race (Other vs. while) is reported here; Test type: Superiority; p = 0.0193, Mixed Models Analysis; Each explanatory variable is reported separately. (Time and intercept estimates are not shown.)
Statistical Analysis 5: Comparison: Radiosurgery/SBRT (Phase III) vs External Beam Radiation Therapy; A general linear mixed-effect model was run with BPI Worst Pain Score (baseline, 3, 6, 12, and 24 months) as the outcome of interest. Age, gender, race, Zubrod performance status, pain medication, tumor type, time, and treatment arm were the covariates considered in each model. Zubrod performance status (0 vs. 1,2) is reported here; Test type: Superiority; p = 0.0016, Mixed Models Analysis; Each explanatory variable is reported separately. (Time and intercept estimates are not shown.)
Statistical Analysis 6: Comparison: Radiosurgery/SBRT (Phase III) vs External Beam Radiation Therapy; A general linear mixed-effect model was run with BPI Worst Pain Score (baseline, 3, 6, 12, and 24 months) as the outcome of interest. Age, gender, race, Zubrod performance status, pain medication, tumor type, time, and treatment arm were the covariates considered in each model. Taking pain medication (No vs. Yes) is reported here; Test type: Superiority; p = 0.0003, Mixed Models Analysis; Each explanatory variable is reported separately. (Time and intercept estimates are not shown.)
Statistical Analysis 7: Comparison: Radiosurgery/SBRT (Phase III) vs External Beam Radiation Therapy; A general linear mixed-effect model was run with BPI Worst Pain Score (baseline, 3, 6, 12, and 24 months) as the outcome of interest. Age, gender, race, Zubrod performance status, pain medication, tumor type, time, and treatment arm were the covariates considered in each model. Tumor type (radioresistant vs. other) is reported here; Test type: Superiority; p = 0.6371, Mixed Models Analysis; Each explanatory variable is reported separately. (Time and intercept estimates are not shown.)

10. Secondary Outcome: Change in EuroQol 5 Dimension (EQ-5D) Index Score Through Two Years (Phase III)
Description: The EQ-5D index score measures health status. Possible scores range from 0 (worst health state) to 1 (best health state), with higher scores indicating better health. Change is calculated as baseline score subtracted from post-baseline score with a positive change indicating improved health status.
Time Frame: Baseline, 3, 6, 12, and 24 months
Population: Questionnaires were not completed by all eligible participants randomized in the phase III component who consented to QOL.. Therefore, the number of participants reported below are the number with the relevant questions answered at baseline and the given time point on each arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Radiosurgery/SBRT (Phase III) | External Beam Radiation Therapy
Number analyzed (Participants) | 152 | 100
score on a scale
  3 months: number analyzed (Participants) | 80 | 53
  3 months | 0.09 (0.19) | 0.09 (0.23)
  6 months: number analyzed (Participants) | 47 | 26
  6 months | 0.08 (0.23) | 0.12 (0.25)
  12 months: number analyzed (Participants) | 39 | 27
  12 months | 0.09 (0.21) | 0.03 (0.25)
  24 months: number analyzed (Participants) | 24 | 12
  24 months | -0.02 (0.26) | -0.02 (0.14)
Statistical Analysis 1: Comparison: Radiosurgery/SBRT (Phase III) vs External Beam Radiation Therapy; A general linear mixed-effect model was run with EQ-5D Index Score (baseline, 3, 6, 12, and 24 months) as the outcome of interest. Age, gender, race, Zubrod performance status, pain medication, tumor type, time, and treatment arm were the covariates considered in each model. Treatment Arm (External Beam Radiation Therapy vs. Radiosurgery/SBRT) is reported here; Test type: Superiority; p = 0.0218, Mixed Models Analysis; Each explanatory variable is reported separately. (Time and intercept estimates are not shown.)
Statistical Analysis 2: Comparison: Radiosurgery/SBRT (Phase III) vs External Beam Radiation Therapy; A general linear mixed-effect model was run with EQ-5D Index Score (baseline, 3, 6, 12, and 24 months) as the outcome of interest. Age, gender, race, Zubrod performance status, pain medication, tumor type, time, and treatment arm were the covariates considered in each model. Age (< 63 years vs. ≥ 63 years) is reported here; Test type: Superiority; p = 0.9437, Mixed Models Analysis; Each explanatory variable is reported separately. (Time and intercept estimates are not shown.)
Statistical Analysis 3: Comparison: Radiosurgery/SBRT (Phase III) vs External Beam Radiation Therapy; A general linear mixed-effect model was run with EQ-5D Index Score (baseline, 3, 6, 12, and 24 months) as the outcome of interest. Age, gender, race, Zubrod performance status, pain medication, tumor type, time, and treatment arm were the covariates considered in each model. Gender (female vs. male) is reported here; Test type: Superiority; p = 0.0696, Mixed Models Analysis; Each explanatory variable is reported separately. (Time and intercept estimates are not shown.)
Statistical Analysis 4: Comparison: Radiosurgery/SBRT (Phase III) vs External Beam Radiation Therapy; A general linear mixed-effect model was run with EQ-5D Index Score (baseline, 3, 6, 12, and 24 months) as the outcome of interest. Age, gender, race, Zubrod performance status, pain medication, tumor type, time, and treatment arm were the covariates considered in each model. Race (Other vs. while) is reported here; Test type: Superiority; p = 0.1140, Mixed Models Analysis; Each explanatory variable is reported separately. (Time and intercept estimates are not shown.)
Statistical Analysis 5: Comparison: Radiosurgery/SBRT (Phase III) vs External Beam Radiation Therapy; A general linear mixed-effect model was run with EQ-5D Index Score (baseline, 3, 6, 12, and 24 months) as the outcome of interest. Age, gender, race, Zubrod performance status, pain medication, tumor type, time, and treatment arm were the covariates considered in each model. Zubrod performance status (0 vs. 1,2) is reported here; Test type: Superiority; p = 0.0003, Mixed Models Analysis; Each explanatory variable is reported separately. (Time and intercept estimates are not shown.)
Statistical Analysis 6: Comparison: Radiosurgery/SBRT (Phase III) vs External Beam Radiation Therapy; A general linear mixed-effect model was run with EQ-5D Index Score (baseline, 3, 6, 12, and 24 months) as the outcome of interest. Age, gender, race, Zubrod performance status, pain medication, tumor type, time, and treatment arm were the covariates considered in each model. Taking pain medication (No vs. Yes) is reported here; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Each explanatory variable is reported separately. (Time and intercept estimates are not shown.)
Statistical Analysis 7: Comparison: Radiosurgery/SBRT (Phase III) vs External Beam Radiation Therapy; A general linear mixed-effect model was run with EQ-5D Index Score (baseline, 3, 6, 12, and 24 months) as the outcome of interest. Age, gender, race, Zubrod performance status, pain medication, tumor type, time, and treatment arm were the covariates considered in each model. Tumor type (radioresistant vs. other) is reported here; Test type: Superiority; p = 0.7732, Mixed Models Analysis; Each explanatory variable is reported separately. (Time and intercept estimates are not shown.)

11. Secondary Outcome: Change in Functional Assessment of Cancer Therapy - General (FACT-G) Total Score Through Two Years (Phase III)
Description: The FACT-G total score gives a combined score of the four domains of health-related quality of life (HRQOL) in cancer patients: Physical, social, emotional, and functional well-being. Possible total scores range from 0 to 108 with higher scores indicating a better HRQOL. Change is calculated as baseline score subtracted from post-baseline score with a positive change indicating improvement in HRQOL.
Time Frame: Baseline, 3, 6, 12, and 24 months
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Radiosurgery/SBRT (Phase III) | External Beam Radiation Therapy
Number analyzed (Participants) | 152 | 100
score on a scale
  3 months: number analyzed (Participants) | 87 | 58
  3 months | 2.4 (16.0) | 5.2 (14.1)
  6 months: number analyzed (Participants) | 50 | 30
  6 months | 5.7 (16.6) | 5.0 (15.8)
  12 months: number analyzed (Participants) | 40 | 28
  12 months | 0.9 (16.6) | 2.9 (20.0)
  24 months: number analyzed (Participants) | 23 | 12
  24 months | -3.8 (16.7) | -2.1 (14.1)
Statistical Analysis 1: Comparison: Radiosurgery/SBRT (Phase III) vs External Beam Radiation Therapy; A general linear mixed-effect model was run with FACT-G total score (baseline, 3, 6, 12, and 24 months) as the outcome of interest. Age, gender, race, Zubrod performance status, pain medication, tumor type, time, and treatment arm were the covariates considered in each model. Treatment Arm (External Beam Radiation Therapy vs. Radiosurgery/SBRT) is reported here; Test type: Superiority; p = 0.5198, Mixed Models Analysis; Each explanatory variable is reported separately. (Time and intercept estimates are not shown.)
Statistical Analysis 2: Comparison: Radiosurgery/SBRT (Phase III) vs External Beam Radiation Therapy; A general linear mixed-effect model was run with FACT-G total score (baseline, 3, 6, 12, and 24 months) as the outcome of interest. Age, gender, race, Zubrod performance status, pain medication, tumor type, time, and treatment arm were the covariates considered in each model. Age (< 63 years vs. ≥ 63 years) is reported here; Test type: Superiority; p = 0.1197, Mixed Models Analysis; Each explanatory variable is reported separately. (Time and intercept estimates are not shown.)
Statistical Analysis 3: Comparison: Radiosurgery/SBRT (Phase III) vs External Beam Radiation Therapy; A general linear mixed-effect model was run with FACT-G total score (baseline, 3, 6, 12, and 24 months) as the outcome of interest. Age, gender, race, Zubrod performance status, pain medication, tumor type, time, and treatment arm were the covariates considered in each model. Gender (female vs. male) is reported here; Test type: Superiority; p = 0.0306, Mixed Models Analysis; Each explanatory variable is reported separately. (Time and intercept estimates are not shown.)
Statistical Analysis 4: Comparison: Radiosurgery/SBRT (Phase III) vs External Beam Radiation Therapy; A general linear mixed-effect model was run with FACT-G total score (baseline, 3, 6, 12, and 24 months) as the outcome of interest. Age, gender, race, Zubrod performance status, pain medication, tumor type, time, and treatment arm were the covariates considered in each model. Race (Other vs. while) is reported here; Test type: Superiority; p = 0.7903, Mixed Models Analysis; Each explanatory variable is reported separately. (Time and intercept estimates are not shown.)
Statistical Analysis 5: Comparison: Radiosurgery/SBRT (Phase III) vs External Beam Radiation Therapy; A general linear mixed-effect model was run with FACT-G total score (baseline, 3, 6, 12, and 24 months) as the outcome of interest. Age, gender, race, Zubrod performance status, pain medication, tumor type, time, and treatment arm were the covariates considered in each model. Zubrod performance status (0 vs. 1,2) is reported here; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Each explanatory variable is reported separately. (Time and intercept estimates are not shown.)
Statistical Analysis 6: Comparison: Radiosurgery/SBRT (Phase III) vs External Beam Radiation Therapy; A general linear mixed-effect model was run with FACT-G total score (baseline, 3, 6, 12, and 24 months) as the outcome of interest. Age, gender, race, Zubrod performance status, pain medication, tumor type, time, and treatment arm were the covariates considered in each model. Taking pain medication (No vs. Yes) is reported here; Test type: Superiority; p = 0.0026, Mixed Models Analysis; Each explanatory variable is reported separately. (Time and intercept estimates are not shown.)
Statistical Analysis 7: Comparison: Radiosurgery/SBRT (Phase III) vs External Beam Radiation Therapy; A general linear mixed-effect model was run with FACT-G total score (baseline, 3, 6, 12, and 24 months) as the outcome of interest. Age, gender, race, Zubrod performance status, pain medication, tumor type, time, and treatment arm were the covariates considered in each model. Tumor type (radioresistant vs. other) is reported here; Test type: Superiority; p = 0.3282, Mixed Models Analysis; Each explanatory variable is reported separately. (Time and intercept estimates are not shown.)

ADVERSE EVENTS:
Time Frame: Collected at 1, 3, 6, 12, and 24 months from randomization.
Description: All-cause mortality reported for all enrolled patients. Adverse events reported for eligible patients who started protocol treatment and have adverse event data. This data was updated when 24 month secondary outcome measures were entered.
Arm/Group | Radiosurgery/SBRT (Phase II) | Radiosurgery/SBRT (Phase III) | External Beam Radiation Therapy
All-Cause Mortality (participants affected / at risk) | 1/46 | 144/217 | 80/136
Serious Adverse Events (participants affected / at risk) | 5/34 | 19/196 | 10/117
Other Adverse Events (participants affected / at risk) | 30/34 | 141/196 | 76/117
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Radiosurgery/SBRT (Phase II) (N=34) | Radiosurgery/SBRT (Phase III) (N=196) | External Beam Radiation Therapy (N=117)
Blood disorder (Blood and lymphatic system disorders) | 0 | 1 | 0
Hemoglobin decreased (Blood and lymphatic system disorders) | 1 | 0 | 2
Pericardial effusion (Cardiac disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1
Duodenal obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1 | 0
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Mucositis oral (Gastrointestinal disorders) | 0 | 1 | 0
Oral pain (Gastrointestinal disorders) | 0 | 1 | 0
Chills (General disorders) | 1 | 1 | 0
Disease progression (General disorders) | 0 | 1 | 0
Fatigue (General disorders) | 0 | 1 | 0
Fever (General disorders) | 2 | 0 | 0
General symptom (General disorders) | 0 | 1 | 0
Catheter related infection [with unknown ANC] (Infections and infestations) | 0 | 0 | 1
Pneumonia [with unknown ANC] (Infections and infestations) | 0 | 1 | 0
Soft tissue infection [with unknown ANC] (Infections and infestations) | 0 | 1 | 0
Stoma site infection [with normal or Grade 1-2 ANC] (Infections and infestations) | 0 | 0 | 1
Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0
Hyperbilirubinemia (Investigations) | 1 | 0 | 0
INR increased (Investigations) | 1 | 0 | 0
Lymphopenia (Investigations) | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 1 | 0
Platelet count decreased (Investigations) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 1 | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 5 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Cognitive disturbance (Nervous system disorders) | 1 | 0 | 0
Ischemia cerebrovascular (Nervous system disorders) | 0 | 0 | 1
Confusion (Psychiatric disorders) | 0 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 3
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Hypotension (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Radiosurgery/SBRT (Phase II) (N=34) | Radiosurgery/SBRT (Phase III) (N=196) | External Beam Radiation Therapy (N=117)
Hemoglobin decreased (Blood and lymphatic system disorders) | 3 | 39 | 16
Abdominal pain (Gastrointestinal disorders) | 0 | 27 | 6
Constipation (Gastrointestinal disorders) | 4 | 32 | 13
Diarrhea (Gastrointestinal disorders) | 0 | 22 | 14
Dysphagia (Gastrointestinal disorders) | 4 | 8 | 1
Nausea (Gastrointestinal disorders) | 5 | 42 | 22
Vomiting (Gastrointestinal disorders) | 1 | 22 | 8
Chest pain (General disorders) | 0 | 12 | 3
Edema limbs (General disorders) | 2 | 22 | 7
Fatigue (General disorders) | 3 | 63 | 31
Fever (General disorders) | 0 | 14 | 6
General symptom (General disorders) | 2 | 6 | 4
Pain [NOS] (General disorders) | 2 | 11 | 6
Pain [other] (General disorders) | 2 | 15 | 12
Fracture (Injury, poisoning and procedural complications) | 0 | 10 | 4
Alanine aminotransferase increased (Investigations) | 1 | 17 | 9
Alkaline phosphatase increased (Investigations) | 3 | 24 | 9
Aspartate aminotransferase increased (Investigations) | 2 | 19 | 10
Creatinine increased (Investigations) | 0 | 10 | 5
Hyperbilirubinemia (Investigations) | 0 | 10 | 5
Leukopenia (Investigations) | 2 | 23 | 8
Lymphopenia (Investigations) | 1 | 20 | 9
Platelet count decreased (Investigations) | 2 | 24 | 9
Weight loss (Investigations) | 1 | 13 | 10
Anorexia (Metabolism and nutrition disorders) | 1 | 28 | 10
Dehydration (Metabolism and nutrition disorders) | 0 | 11 | 2
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 32 | 12
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 30 | 8
Hypocalcemia (Metabolism and nutrition disorders) | 2 | 29 | 10
Hypokalemia (Metabolism and nutrition disorders) | 2 | 17 | 9
Hyponatremia (Metabolism and nutrition disorders) | 2 | 17 | 8
Back pain (Musculoskeletal and connective tissue disorders) | 14 | 60 | 30
Bone pain (Musculoskeletal and connective tissue disorders) | 5 | 7 | 7
Joint pain (Musculoskeletal and connective tissue disorders) | 2 | 16 | 3
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 23 | 7
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 | 12 | 3
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 2 | 11 | 4
Neck pain (Musculoskeletal and connective tissue disorders) | 3 | 13 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 24 | 12
Dizziness (Nervous system disorders) | 0 | 13 | 4
Headache (Nervous system disorders) | 3 | 12 | 5
Peripheral motor neuropathy (Nervous system disorders) | 2 | 4 | 3
Peripheral sensory neuropathy (Nervous system disorders) | 6 | 17 | 8
Anxiety (Psychiatric disorders) | 1 | 11 | 3
Confusion (Psychiatric disorders) | 0 | 10 | 8
Urinary retention (Renal and urinary disorders) | 2 | 0 | 4
Urogenital disorder (Renal and urinary disorders) | 1 | 11 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 17 | 12
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 32 | 12
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 10 | 4
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 10 | 6
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 1 | 1
Rash desquamating (Skin and subcutaneous tissue disorders) | 2 | 6 | 3
Hypotension (Vascular disorders) | 2 | 13 | 1
Thrombosis (Vascular disorders) | 1 | 13 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI's are required to abide by the sponsor's publication guidelines which require review by coauthors and subsequent review and approval by the sponsor

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-23): https://cdn.clinicaltrials.gov/large-docs/74/NCT00922974/Prot_SAP_000.pdf